CLINICAL TRIAL: NCT03044314
Title: Outpatient Vasodilator Assessment Using Iloprost in Pulmonary Hypertension (The OVATION Study)
Brief Title: Outpatient Vasodilator Assessment Using Iloprost in Pulmonary Hypertension
Acronym: OVATION
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Duke University (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00075840
Record Dates: First submitted 2016-10-06; First posted 2017-02-07 (Estimated); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; vasodilator challenge; echocardiography; outcomes; iloprost; inhaled nitric oxide
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Iloprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Iloprost and nitric oxide administration (Experimental): Each patient will receive 40 ppm inhaled nitric oxide and 2.5-5 mcg inhaled iloprost in the catheterization laboratory with assessment of hemodynamic response. Patients will also receive 2.5-5 mcg iloprost during echocardiographic assessment.
  Interventions: Drug: Iloprost and nitric oxide administration

INTERVENTIONS:
Drug: Iloprost and nitric oxide administration — Iloprost will be administered by the I-neb ultrasonic nebulizer (Respironics, Cedar Grove, New Jersey) with a disposable attachment that allows for administration to a supine patient at a concentration of 10 µg/ml with a 10 minute dose of 2.5 µg and then repeated to a cumulative dose of 5.0 µg if tolerated.
  Other Names: Ventavis

SUMMARY:
This study will compare the clinical efficacy of inhaled iloprost as an invasive, selective vasodilator in the cardiac catheterization laboratory in patients with pulmonary hypertension to the gold standard of inhaled nitric oxide. It will also examine whether echocardiographic estimates of response to inhaled iloprost can predict responsiveness to invasive vasodilator testing in patients with pulmonary hypertension.

DETAILED DESCRIPTION:
Iloprost was the first inhaled prostacyclin analogue to be FDA-approved for the treatment of pulmonary arterial hypertension. Iloprost aerosol has been shown to significantly improve pulmonary hemodynamics in patients with idiopathic pulmonary hypertension (PH), with an effect greater than nitric oxide and sildenafil. It has also been shown to be more effective than nitric oxide at reducing pulmonary arterial pressure (PAP) than prostacyclin infusion when used in the cardiac catheterization laboratory. Because of its administration through inhalational means, iloprost has the advantage of selective action on the pulmonary vasculature with avoidance of the systemic side effects that plague many of the other treatments for PH. The investigators intend to compare the efficacy of inhaled iloprost in reducing pulmonary artery pressure to the gold standard of nitric oxide in patients with pulmonary hypertension.

Without an established noninvasive algorithm to identify beneficial hemodynamic response to vasodilators, patients with pulmonary hypertension (PH) are routinely subjected to expensive and invasive testing. Echocardiography is routinely used to facilitate a diagnosis of PH and a few echocardiographically-derived estimates have even been shown to correlate with vasodilator responsiveness and survival. Dynamic, real time changes in echocardiographic parameters have not been previously evaluated as a predictor of vasodilator responsiveness or of clinical outcome. The investigators will examine whether echocardiographic changes in response to inhaled iloprost can predict invasively derived vasodilator responsiveness and help assess prognosis in patients with pulmonary hypertension, possibly even obviating the need for invasive testing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients no younger than 18 years of age
* Recently diagnosed pulmonary hypertension (defined by RV systolic pressure of ≥ 40 mmHg as measured by echocardiography), going for invasive hemodynamic assessment for pulmonary hypertension
* Normal left ventricular function defined as a left ventricular ejection fraction (LVEF) greater than or equal to 50%

Exclusion Criteria:

* Heart failure (LVEF < 50%, diastolic dysfunction > stage 1, history or symptoms of left heart failure) - Group II pulmonary hypertension
* 2+ or higher MR or AI
* Inadequate echocardiographic windows
* Pregnancy
* Systolic blood pressure ≤ 90 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2020-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Krasuski, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were identified from pulmonary hypertension clinic as well as those referred to the catheterization lab for their initial diagnostic right heart catheterization for evaluation of pulmonary hypertension.
Groups:
- Nitric Oxide and Iloprost Administration: Each patient will receive 40 ppm inhaled nitric oxide and 2.5-5 mcg inhaled iloprost in the catheterization laboratory with assessment of hemodynamic response. Patients will also receive 2.5-5 mcg iloprost during echocardiographic assessment.
  Iloprost and nitric oxide administration: Iloprost will be administered by the I-neb ultrasonic nebulizer (Respironics, Cedar Grove, New Jersey) with a disposable attachment that allows for administration to a supine patient at a concentration of 10 µg/ml with a 10 minute dose of 2.5 µg and then repeated to a cumulative dose of 5.0 µg if tolerated.
Period: Overall Study
Arm/Group | Nitric Oxide and Iloprost Administration
Started | 27
Completed | 23
Not Completed | 4
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1
Not completed — Connector tubing not available | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Arm/Group | Nitric Oxide and Iloprost Administration
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Invasively Measured Pulmonary Artery Pressures After Challenge With iNO (Inhaled Nitrous Oxide) and Iloprost
Time Frame: Baseline and approximately 30 minutes
Population: Participants who completed the study. Each participant was analyzed after challenge with iNO and after challenge with iloprost.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Inhaled Nitric Oxide; Iloprost: Each patient will receive 40 ppm inhaled nitric oxide and 2.5-5 mcg inhaled iloprost in the catheterization laboratory with assessment of hemodynamic response. Patients will also receive 2.5-5 mcg iloprost during echocardiographic assessment.
  Iloprost and nitric oxide administration: Iloprost will be administered by the I-neb ultrasonic nebulizer (Respironics, Cedar Grove, New Jersey) with a disposable attachment that allows for administration to a supine patient at a concentration of 10 µg/ml with a 10 minute dose of 2.5 µg and then repeated to a cumulative dose of 5.0 µg if tolerated.
Arm/Group | Inhaled Nitric Oxide | Iloprost
Number analyzed (Participants) | 23 | 23
percent change | 10.7 (7.1) | 13.3 (12.5)
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide vs Iloprost; Null hypothesis: inhalation with iNO (the gold standard) would provide greater response than the comparator (iloprost); Test type: Superiority; p = 0.148, t-test, 2 sided

2. Secondary Outcome: Percent Change in Systolic Pulmonary Arterial Pressure After Vasodilator Challenge
Time Frame: Baseline and during vasodilator inhalation, approximately 30 minutes
Population: Participants who completed the study. Two patients refused to undergo echocardiography and repeat inhalation of iloprost.
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- Inhaled Nitric Oxide and Iloprost Administration: Each patient will receive 40 ppm inhaled nitric oxide and 2.5-5 mcg inhaled iloprost in the catheterization laboratory with assessment of hemodynamic response. Patients will also receive 2.5-5 mcg iloprost during echocardiographic assessment.
  Iloprost and nitric oxide administration: Iloprost will be administered by the I-neb ultrasonic nebulizer (Respironics, Cedar Grove, New Jersey) with a disposable attachment that allows for administration to a supine patient at a concentration of 10 µg/ml with a 10 minute dose of 2.5 µg and then repeated to a cumulative dose of 5.0 µg if tolerated.
Arm/Group | Inhaled Nitric Oxide and Iloprost Administration
Number analyzed (Participants) | 21
percentage of change | 0 (0)

3. Secondary Outcome: Number of Participants Who Respond After Vasodilator Challenge
Description: Dichotomize the vasodilator response into responders and nonresponders, based on a 10 mmHg drop in PA pressure and a mean pressure <40mmHg determined invasively. Receiver operating characteristic (ROC) curves will evaluate the echocardiographic parameters for prediction of vasodilator response.
Time Frame: Baseline and during vasodilator inhalation, approximately 30 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide | Iloprost
Number analyzed (Participants) | 23 | 23
Participants | 1 | 4
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide vs Iloprost; Null hypothesis was that fewer patients receiving iloprost (new agent) would respond compared to iNO (the gold standard); Test type: Superiority; p = 0.346, Fisher Exact

4. Secondary Outcome: Number of Participants With Clinical Response to Vasodilator Challenge by Echo
Description: Measure the clinical response to vasodilator challenge during echocardiography, by tracking the changes of echo parameters (such as RVSP) before and after iloprost challenge, as well as through the 3 and 12 month follow-up visits.
Time Frame: Baseline, approximately 30 minutes, 3 months, and 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide and Iloprost Administration
Number analyzed (Participants) | 21
Participants
  Baseline | 0
  30 minutes | 0
  3 months | 0
  12 months | 0

5. Secondary Outcome: Association of Change in Pressures After Vasodilator Challenge With Clinical Outcomes
Description: Observe the association of the percent change of echocardiographically estimated pressures after iloprost challenge with mid-term clinical outcomes (all cause mortality and all cause mortality +/- hospitalization). These data will be collected at 3 months and at 12 months. Data from all hospitalizations will be collected though we will make special note of those related to pulmonary hypertension.
Time Frame: 3 months and 12 months
Population: 0 participants had a change of echocardiographically estimated pressures, as indicated in outcome #4
Arm/Group | Inhaled Nitric Oxide and Iloprost Administration
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Inhalation of iNO for 5 minutes with immediate off-effect when stopped. Inhalation of iloprost for 30 minutes and 20-30 minute half-life (negligible effect at 2 hours). Patients observed for hypotension, dizziness, cough, bleeding, etc. All patients observed in the cath lab and holding area after inhalation for >2 hours post-administration. Questioned about symptoms prior to discharge. Mid-term clinical outcome data will be collected at 3 months and at 12 months.
Groups:
- Iloprost and Nitric Oxide Administration: Each patient will receive 40 ppm inhaled nitric oxide and 2.5-5 mcg inhaled iloprost in the catheterization laboratory with assessment of hemodynamic response. Patients will also receive 2.5-5 mcg iloprost during echocardiographic assessment.
  Illoprost and nitric oxide administration: Iloprost will be administered by the I-neb ultrasonic nebulizer (Respironics, Cedar Grove, New Jersey) with a disposable attachment that allows for administration to a supine patient at a concentration of 10 µg/ml with a 10 minute dose of 2.5 µg and then repeated to a cumulative dose of 5.0 µg if tolerated.
Arm/Group | Iloprost and Nitric Oxide Administration
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT03044314/Prot_SAP_000.pdf